CLINICAL TRIAL: NCT02883920
Title: Work-related Respiratory Symptoms in Champagne Vineyard Workers
Acronym: VIN-ALLERGO
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2015Ao004
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Respiratory Symptoms
MeSH Terms: conditions — Signs and Symptoms, Respiratory | interventions — Sensitivity and Specificity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- workers of Champagne vineyard
  Interventions: Other: Allergy and respiratory functional tests

INTERVENTIONS:
Other: Allergy and respiratory functional tests

SUMMARY:
Work related asthma and rhinitis are frequent diseases with a significant morbidity and a social and economic impact. Farmers are highly exposed to various inhaled agents such as organic or inorganic dust, endotoxin, micro-organisms, pollen, mites, moulds, animal danders and pesticides, inducing rhinitis, asthma, chronic bronchitis, hypersensitivity pneumonitis and organic dust toxic syndrome. Work related respiratory symptoms are frequent in crop farmers. Allergic rhinitis and respiratory symptoms in fruit farmers are mainly related to pollen allergy, especially gramineae pollen. They can also be related to the use of pesticides or exposure to mites .

DETAILED DESCRIPTION:
Aim of the study were :

to determine the prevalence of work related respiratory symptoms in workers of Champagne vineyard in France to analyze the relationships between respiratory symptoms, occupational exposure and sensitization profile in workers of Champagne vineyard in France

ELIGIBILITY:
Inclusion Criteria:

* workers of Champagne vineyard
* aged > 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: workers of Champagne vineyard.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Sensitization | Day 0
  A positive skin prick test was defined as the presence of a mean wheal diameter of 3 mm or more than the negative control. Sensitization was defined by a positive skin reaction to one or more allergens

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France

REFERENCES:
- [Background] Perotin JM, Barbe C, Nguyen KL, Fontaine JF, Gabignon Y, Nardi J, Launois C, Lebargy F, Lavaud F, Deslee G. Work-related respiratory symptoms in Champagne vineyard workers. Eur Ann Allergy Clin Immunol. 2015 Sep;47(5):140-4. PMID 26356997